CLINICAL TRIAL: NCT05274490
Title: Chronic Obstructive Pulmonary Disease Prognosis in Sars-covid 2 Infection
Brief Title: COPD Prognosis in Covid Patients
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Islam Mokhtar Ahmed, lecturer of anesthesia and intensive care, Sohag University
Other Study IDs: soh-Med-22-1-26
Record Dates: First submitted 2022-03-05; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Respiratory Failure
Keywords: copd, prognosis, covid
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive | interventions — Intubation; Respiration, Artificial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- copd patients with covid infection
  Interventions: Procedure: intubation and mechanical ventilation
- non-copd patients with covid infection
  Interventions: Procedure: intubation and mechanical ventilation

INTERVENTIONS:
Procedure: intubation and mechanical ventilation — patients who were in need were intubated and mechanically ventilated

SUMMARY:
In this prospective observational study, patients were selected from attendees of the intensive care unit. Different measures and outcomes had been studied and compared between patients with and without COPD, including hospitalization, medical costs, length of Intensive care stay, respiratory failure, and death rate.

ELIGIBILITY:
Inclusion Criteria:

* Age: more than 20 years old.

  * Both Males and females will be included.
  * COPD patients.
  * Recent confirmed the diagnosis with SARS-COV-2.

Exclusion Criteria:

* Pregnancy.

  * Malignancy.
  * Immunodeficiency disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male or female patient more than 20 years old, recently diagnosed covid positive
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
SOFA score measurement in both groups | 2 weeks
  monitoring of SOFA items along two weeks

SECONDARY OUTCOMES:
prognosis of the disease | 2 weeks
  hospital stay, nedd for mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt